CLINICAL TRIAL: NCT01914861
Title: Cortisol Diurnal Variation and the Risk for Developing Post Traumatic Stress Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: Sheba-0361-13-AJW-CTIL
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Posttraumatic Stress Disorders; Cortisol Diurnal Variation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma cortisol levels plasma neuropeptide y

GROUPS / COHORTS (1):
- Men/Women, 21-65, following exposure to a traumatice event

SUMMARY:
The purpose of this study is to examine a possible link between the time of day of exposure to a traumatic event and the risk of developing post-traumatic stress disorder. Clinical and biological correlates will also be examined from this perspective.

ELIGIBILITY:
Inclusion Criteria:

1. Persons 21-65 years old, who have been exposed to an event meeting the following DSM-IV criterion for Acute Stress Disorder:

   Criteria A.1 and A.2 At least one of Criteria B1-5A.1
2. Who provide written, informed consent to participate in the study.

Exclusion Criteria:

1. Physical injury that would contraindicate participation or interfere with a subject's ability to give informed consent or cooperate with the screening or collection of initial measures. Examples include severe burn injury, life-threatening medical or surgical condition, condition requiring surgical intervention under general anesthesia, as indicated by Abbreviated Injury Scale (AIS), or by clinical judgment;
2. Head injury involving confusion, loss of consciousness, or amnesia;
3. Medical conditions such as extreme obesity, psoriasis, herpes, Cushing's syndrome, current infectious disease, current viral disease, tuberculosis, unstable diabetes or hypertension, myasthenia gravis, and heart failure. Persons taking medications that can interfere with the HPA axis (e.g.,steroids, betablockers,indomethacin) will be excluded;
4. Weight below 45 or above 120 kg.
5. Pregnancy (in suggestive cases, a pregnancy test will be performed);
6. Traumatic exposure that reflects ongoing victimization (e.g., domestic violence) to which the subject is likely to be re-exposed during the study period.
7. Overt psychopathology, intoxication, or under the influence of substances.
8. Evidence or history of schizophrenia, bipolar, other psychotic condition;
9. Prior history of PTSD;
10. Current or past history of dementia, amnesia, or other cognitive disorder predating trauma exposure;
11. Assessed serious suicide risk. -

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men/Women, age 21-65, who have arrived at the Chaim Sheba Medical Center ER within six hours of exposure to a traumatic event.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Development of Posttraumatic stress disorder | six months

SECONDARY OUTCOMES:
Biological correlates of post-traumatic stress disorder | six months
correlation between development of Posttraumatice stress disorder and time of traumatic event | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel